CLINICAL TRIAL: NCT05130996
Title: Observational Study Evaluating Safety and Performance of Dental Implant Systems (5 Implant Ranges: IDAll, IDBio, IDCam, IDMax, ID3; 3 Types of Prosthetic Parts: Sealed, Screw-retained and Removable) in Subjects Followed During 18 Month
Brief Title: Observational Study Evaluating Safety and Performance of IDI Dental Implant Systems in Subjects Followed for 18 Months.
Status: Recruiting | Type: Observational
Sponsor: Implants Diffusion International (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A02389-48
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dental Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: dental prothesis — 5 ranges of implants can be used : IDAll, IDBio, IDCam, IDMax, ID3

SUMMARY:
Post-Market Clinical Follow-Up to evaluate the safety and performance of IDI dental implant systems : confirmation of osseointegration of the different implants at the loading visit (between 2 and 6 months after surgery).

DETAILED DESCRIPTION:
The aim of the present study is to carry out post-marketing clinical monitoring of the medical device used in accordance with the instructions for use according to a medical strategy intended for the person who is suitable for this research which is not fixed in advance by an investigation plan and is part of the current practice of the surgeon.

This is a comparative, prospective, multicenter observational study

The osteointegration reached between 2 and 6 months after surgery will be evaluated by clinical and radiological examinations:

ELIGIBILITY:
Inclusion Criteria:

* Subject receiving an insertion of an aesthetic and functional oral prosthesis on IDI implant systems (IDAll, IDBio, IDCam, IDMax or ID3) for at least one of the following indications:

  * Single, partial or complete edentulousness
  * Stabilization of a removable prosthesis
* Subject having received an information sheet on the study and having indicated their non-objection before starting the procedures specific to the protocol.
* ASA score (American Society of Anesthesiologists) <3.
* If a recent extraction has been performed at the site of the implantation area, the healing period should be at least 2 months.
* Sufficient bone volume (minimum 4mm) to accommodate dental implants.

Exclusion Criteria:

* Pregnant or breastfeeding woman.
* Inability of the subject to maintain reasonable oral hygiene in accordance with study requirements.
* Parafunctional habits, such as bruxism or temporomandibular joint disease.
* Different pathologies of the oral mucosa such as: benign mucous pemphigoid, desquamative gingivitis, malignant tumor of the oral cavity, bolus erosive diseases of the oral mucosa.
* Disorders of bone metabolism.
* Untreated, unmanaged caries and / or periodontal disease.
* Need for simultaneous bone grafting and / or sinus lift in the intended implant area.
* Medical history making insertion of the implant unfavorable.
* Lack of cooperation. Subject may not comply with study procedures.
* Heavy use of tobacco (more than 10 cigarettes per day), drugs and / or alcohol.
* Treatment with bisphosphonates, steroids or anticonvulsants.
* Unbalanced diabetes.
* Subject receiving radiotherapy, chemotherapy or any other immunosuppressive treatment. Subjects who received radiation therapy to the head and neck area at any time should not be included.
* Congenital or acquired (HIV positive) diseases that compromise the immune system.
* Uncontrolled bleeding disorders such as: haemophilia, thrombocytopenia, granulocytopenia.
* Renal failure.
* Organ transplant recipient.
* Malignant diseases.
* Psychotic illnesses.
* Hypersensitivity to one of the components of the implant in general and to titanium in particular. It is the surgeon's responsibility to ensure that the subject does not have known allergies to any of the components of the material listed on the product label.
* Sports or physical activities including violent shocks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult population receiving an IDI implant under the conditions of use intended by the manufacturer.
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Osteointegration achieved between 2 and 6 months evaluated by clinical examination | between 2 and 6 months after the surgery (dental implantation)
  Measurement of the stability index of the implant with OSSEO100
Osteointegration achieved between 2 and 6 months evaluated by radiological examination | between 2 and 6 months after the surgery (dental implantation)
  Measurement of the bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Office, Paris, France

IPD SHARING:
Plan to Share IPD: No